CLINICAL TRIAL: NCT02593396
Title: A Randomized, Double-Blind, Parallel-Group, Placebo-Controlled Trial Of Bupropion Hydrochloride Sustained-Release In The Treatment Of Sexual Dysfunction In Men On Methadone Maintenance Therapy
Brief Title: Bupropion in Sexual Dysfunction Among Methadone Maintenance Treatment Men
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: University of Malaya (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: AY001
Record Dates: First submitted 2015-10-05; First posted 2015-11-02 (Estimated); Results first posted 2019-07-12 (Actual); Last update posted 2019-08-01 (Actual); Status verified 2019-07

CONDITIONS: Sexual Dysfunctions, Psychological; Hypoactive Sexual Desire Disorder; Erectile Dysfunctions
Keywords: sexual dysfunctions; erectile dysfunctions; hypoactive sexual desire dysfunctions
MeSH Terms: conditions — Sexual Dysfunctions, Psychological; Erectile Dysfunction | interventions — Bupropion

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- placebo (Placebo Comparator): Placebo BD
  Interventions: Drug: placebo
- Active (Experimental): Bupropion hydrochloride sustained-release 150mg BD
  Interventions: Drug: Bupropion hydrochloride sustained-release

INTERVENTIONS:
Drug: Bupropion hydrochloride sustained-release — Up to 70 eligible patients will be randomly assigned to Bupropion Hydrochloride Sustained-Release or placebo treatment groups in a 1:1 ratio using a computer-generated table of random numbers through the use of the Randomization.com program. Subjects will be randomized to to Bupropion Hydrochloride Sustained-Release 150mg b.d. (n = 35) or placebo b.d (n = 35)The study drug will be repacked in the standard capsules by the research assistant who is not involved in the assessment of the study. The study drug and placebo will be packaged in sets of 11 (1 tablet per day for 3 days, followed by 2 tablets per day for 4 days.) for the first week. Subsequently, the study drug and placebo will be packaged in sets of 14 (2 tablets per day for 7 days.).
  Other Names: wellbutrin SR
  Arms: Active
Drug: placebo — Up to 70 eligible patients will be randomly assigned to Bupropion Hydrochloride Sustained-Release or placebo treatment groups in a 1:1 ratio using a computer-generated table of random numbers through the use of the Randomization.com program. Subjects will be randomized to to Bupropion Hydrochloride Sustained-Release 150mg b.d. (n = 35) or placebo b.d (n = 35)
  Arms: placebo

SUMMARY:
The purpose of this study is to assess the tolerability, safety, and efficacy of bupropion hydrochloride sustained-release in the treatment of sexual dysfunction in men on methadone maintenance therapy.

DETAILED DESCRIPTION:
This is a single-center (University Malaya Medical Centre), randomized, double-Blind, placebo-controlled versus bupropion hydrochloride sustained-releases study trial on 70 men who have methadone emergent sexual dysfunction. Bupropion hydrochloride sustained-release (Wellbutrin SR) 150mg once a day for 7 days then 150mg twice a day for 42 days. Taken orally by the subjects.The total duration of the study is expected to be 24 months. 20months for subject recruitment and 4 months for final subject follow-up.

The primary endpoint is Mean improvement in scores on the Clinical Global Impression Scale adapted for sexual Function (CGI-SF). Secondary endpoints are Change from baseline International Index of Erectile Function (IIEF-15) score. Mean improvement in scores on the sexual desire inventory 2 (SDI2). Other evaluation included: Montgomery-Åsberg Depression Rating Scale (MADRS- Malay version ), Mini International Neuropsychiatric Interview (M.I.N.I), Opiate Treatment Index (OTI), World health organization Quality of Life-Brief Scale (WHOQoL-Brief, Malay version), Malay Version of the Golombok-Rust Inventory of Marital State (Mal-GRIMS) and Rapid urine drug test. Safety evaluation included: Incidence of adverse events. Data will be analyzed using linear mixed-effects model.

ELIGIBILITY:
Inclusion Criteria:

* Had a diagnosis of opioid dependence base on Diagnostic and Statistical Manual of Mental Disorders, Fourth Edition (DSM-IV) criteria
* While taking a stable dose of methadone In UMMC (University Malaya Medica Centre) and University Malaya centre of Addiction Science (UMCAS) outpatient clinic for ≥ 6 months
* Were experiencing constant sexual dysfunction for ≥ 4 weeks
* Were in a stable sexual relationship with a female partner for ≥ 6 months

Exclusion Criteria:

* Severe behavior disturbances or psychotic symptoms
* Obvious organic illnesses caused the sexual dysfunction (such as diabetics or patients with heart and vascular disease)
* Those with history of sexual dysfunction before methadone therapy
* Receiving antiviral treatment for viral hepatitis or HIV, or androgen replacement treatment.
* History of an eating disorder (eg, anorexia, bulimia) or seizures (eg, epilepsy)
* Using other psychotropic medications other than methadone
* Clinical significant abnormal laboratory values.
* Clinically significant abnormal ECG. Documented history of other psychiatric diagnosis (schizophrenia, bipolar disorder, major depressive disorder, organic brain disorder, dementia etc.)
* Refused to give participate.

Ages: 18 Years to 65 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 80 (Actual)
Dates: Start 2015-12 (Actual); Primary Completion 2017-12 (Actual); Study Completion 2017-12 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Anne Yee, Principal Investigator — University Malaya Medical Center
Locations (1):
- University Malaya Medical Center, Kuala Lumpur, Selangor, Malaysia

RESULTS

PARTICIPANT FLOW:
Recruitment Details: All the male subjects who attended the methadone maintenance clinic from December 2015 to December 2017 in University Malaya Medical Center (UMMC) and University Malaya Center of Addiction Science Studies (UMCAS) were approached.Screening data was reviewed to determine subject eligibility.
Pre-assignment Details: This study screened 109 and included 80 (73.4%) male patients who met all inclusion criteria and none of the exclusion criteria.
Period: Overall Study
Arm/Group | Placebo | Active
Started | 40 | 40
At Least Done One Efficacy Assessment (At least one efficacy assessment after the baseline visit.) | 36 | 36
Completed | 25 | 26
Not Completed | 15 | 14

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Placebo | Active | Total
Number analyzed (Participants) | 40 | 40 | 80
Age, Continuous [Mean (Standard Deviation); unit: years] | 43.50 (10.09) | 42.30 (9.49) | 42.83 (9.68)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 0 | 0 | 0
  Male | 40 | 40 | 80
Race/Ethnicity, Customized [Count of Participants; unit: Participants]
  Race: Malay | 34 | 34 | 68
  Race: Chinese | 5 | 3 | 8
  Race: Indian | 1 | 1 | 2
  Race: Others | 0 | 2 | 2
Malay version of International Index of Erectile Function (Mal-IIEF-15) [Mean (Standard Deviation); unit: units on a scale] — Mal-IIEF-15 is a 15-item, multi-dimensional self-reporting instrument for the evaluation of male sexual function for the past 4 weeks. Items 1-10 is 6-point Likert-type scale from '0' (= No sexual activity) to '5' (= Almost always or always). Items 11-15 is 5-point Likert-type scale from '1' (= Almost never or never) to '5 '(= 'Almost always or always').The total Mal-IIEF-15 range from 5 (minimum) to 75 (Maximum). The higher score reflecting a better sexual function.
  units on a scale | 42.44 (16.43) | 41.80 (19.13) | 42.12 (17.78)
Total Malay version of the SDI-2 (SDI-2-BM) [Mean (Standard Deviation); unit: units on a scale] — This scale contains 14 items which yield two domain scores: dyadic sexual desire (DSD) and solitary sexual desire (SSD). Items 1,2, 10 are 8-point Likert scale from '0' (= not at all) to '7' (= more than once a day) concerning frequency of desire. Remaining Items are 9-point Likert scale from '0' (= 'no desire') to '8' (= 'strong desire'). DSD has 8 items and SSD has 3 items. The total sores for DSD range from 0 to 62, and SSD, range from 0 to 23. All items are summed up to dictate the total sexual desire (total score = 0 to 109). Higher scores reflect higher sexual desire.
  units on a scale | 42.87 (15.83) | 42.58 (14.97) | 42.73 (15.4)

OUTCOME MEASURES:

1. Primary Outcome: Number of Participants With a Score of ≤2 (Much/Very Much Improved) on the Clinical Global Impression Scale Adapted for Sexual Function (CGI-SF) at Week 6 Between Placebo and Active Group
Description: This scale assesses the changes of the sexual function. Scores range from 1 (normal/very much improved) to 7 (most extreme sexual dysfunction/very much worse). Lower scores indicate better sexual functioning.
Time Frame: assessed at baseline, day 14(week 2), day 28(week four) and day 42 (week 6), data at day 42 (week 6) reported
Population: Intention-to-treat (ITT) analyses were used for all efficacy variables and included all patients who had been randomized, took at least 1 dose of study trial medication and had at least one efficacy assessment after the baseline visit. There were four patients in each arm did not come for first efficacy assessment, Hence, excluded from analysis.
Measure: Count of Participants; unit: Participants
Arm/Group | Placebo | Active
Number analyzed (Participants) | 36 | 36
Participants | 10 | 21

2. Secondary Outcome: Mean Difference of Malay Version of International Index of Erectile Function (Mal-IIEF-15) at Week 6 Between Placebo and Active Group
Description: Mal-IIEF-15 is a 15-item, multi-dimensional self-reporting instrument for the evaluation of male sexual function for the past 4 weeks, consisted of five domains; 1) Erectile Function: sum of items 1, 2, 3, 4, 5 & 15. Total score range =1-30. 2) Orgasmic Function: sum of items 9 and 10. Total score range = 0 -10. 3) Sexual Desire: sum of items 11 and 12. Total score range = 2 -10. 4) Intercourse Satisfaction : sum of scores for Questions 6, 7 and 8. Total score range = 0 -15. 5) Overall Satisfaction: sum of items 13 and 14.Total score range = 2 -10. Items 1-10 is 6-point Likert-type scale from '0' (= No sexual activity) to '5' (= Almost always or always). Items 11-15 is 5-point Likert-type scale from '1' (= Almost never or never) to '5 '(= 'Almost always or always').The total Mal-IIEF-15 range from 5 (minimum) to 75 (Maximum). Higher score indicates better outcome in all domain.
Time Frame: assessed at baseline, day 14(week 2), day 28(week four) and day 42 (week 6), data at day 42 (week 6) reported
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Placebo | Active
Number analyzed (Participants) | 36 | 36
score on a scale
  IIEF total | 43.81 (19.86) | 52.53 (16.14)
  Mal-IIEF-15, Erectile function domain | 18.06 (9.43) | 22.56 (7.69)
  Mal-IIEF-15, Orgasmic function domain | 5.99 (3.75) | 7.30 (2.92)
  Mal-IIEF-15, Sexual desire domain | 6.04 (1.97) | 6.77 (1.91)
  Mal-IIEF-15, Intercourse satisfaction domain | 6.46 (4.18) | 8.78 (3.77)
  Mal-IIEF-15, Overall satisfaction domain | 7.14 (2.41) | 7.10 (2.29)

3. Secondary Outcome: Mean Difference of Malay Version of Sexual Desire Inventory 2 (SDI-2) Score at Weeks 6 Between Placebo and Active Groups
Description: This scale contains 14 items which yield two domain scores: dyadic sexual desire (DSD) and solitary sexual desire (SSD). Items 1,2, 10, 14 are 8-point Likert scale from '0' (= not at all) to '7' (= more than once a day) concerning frequency of desire. Remaining Items are 9-point Likert scale from '0' (= 'no desire') to '8' (= 'strong desire'). DSD has 8 items and SSD has 3 items. The total sores for DSD range from 0 to 62, and SSD, range from 0 to 23. All items are summed up to dictate the total sexual desire (total score = 0 to 112). Higher scores reflect higher sexual desire.
Time Frame: Assessed at baseline, day 14(week 2), day 28(week four) and day 42 (week 6), data at day 42 (week 6) reported
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Placebo | Active
Number analyzed (Participants) | 36 | 36
score on a scale
  SDI-2 | 47.36 (21.09) | 53.53 (15.88)
  DSD | 29.99 (13.44) | 36.08 (10.17)
  SSD | 6.87 (5.97) | 7.45 (4.97)

ADVERSE EVENTS:
Time Frame: 6 weeks
Description: patient self-report
Arm/Group | Placebo | Active
All-Cause Mortality (participants affected / at risk) | 0/36 | 0/36
Serious Adverse Events (participants affected / at risk) | 0/36 | 0/36
Other Adverse Events (participants affected / at risk) | 8/36 | 13/36
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Placebo (N=36) | Active (N=36)
Insomnia (General disorders) | 1 (1) | 6 (6) — Insomnia
skin rash (Skin and subcutaneous tissue disorders) | 0 (0) | 3 (3)
inability to concentrate (Psychiatric disorders) | 0 (0) | 2 (2)
constipation (Gastrointestinal disorders) | 2 (2) | 2 (2)
nausea (Gastrointestinal disorders) | 2 (2) | 0 (0)
ineffectiveness (General disorders) | 3 (3) | 0 (0)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes; Agreement restricts PI disclosure of results: Yes; Restriction type: embargo of 60 days or less

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2015-03-01): https://cdn.clinicaltrials.gov/large-docs/96/NCT02593396/Prot_SAP_000.pdf